CLINICAL TRIAL: NCT07074509
Title: Comparative Study of Effectiveness of Manual Therapy and Extracoropral Shock Wave Therapy in Patients With Carpal Tunnel Syndrome
Brief Title: Effectiveness of Manual Therapy and Extracoropral Shock Wave Therapy in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Naser Elsayed Elderby, Resident of Rheumatology, Rehabilitation and Physical Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36208/12/22
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Manual Therapy; Extracoropral Shock Wave Therapy; Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Musculoskeletal Manipulations; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Patients were treated by manual therapy in the form of nerve gliding, soft tissue release, and carpal bone mobilization, three sessions per week for 4weeks.
  Interventions: Other: Manual therapy
- Group 2 (Experimental): Patients were treated by extracorporeal shock wave therapy. 4 sessions, one week apart, 2000 pulses per session, intensity 1.6 mj/mm, and frequency 8Hz.
  Interventions: Other: Extracorporeal shock wave therapy

INTERVENTIONS:
Other: Manual therapy — Patients were treated by manual therapy in the form of nerve gliding, soft tissue release, and carpal bone mobilization, three sessions per week for 4weeks.
  Arms: Group 1
Other: Extracorporeal shock wave therapy — Patients were treated by extracorporeal shock wave therapy. 4 sessions, one week apart, 2000 pulses per session, intensity 1.6 mj/mm, and frequency 8Hz.
  Arms: Group 2

SUMMARY:
This study aimed to compare the effectiveness of manual therapy and extracorporeal shock wave therapy in patients with mild to moderate carpal tunnel syndrome.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS), the most common peripheral neuropathy in the upper limb, occurs due to the entrapment of the median nerve at the wrist. Treatment options for CTS consist of wrist splints, physical modalities, local corticosteroid injections, and surgical release.

Extracorporeal shockwave therapy (ESWT) is a noninvasive technique that uses single-pulse acoustic waves. These pulses are generated outside the body and focused on a specific part of the body.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes.
* Patients with mild and moderate carpal tunnel syndrome (CTS).

Exclusion Criteria:

* Severe cases of CTS.
* History of carpal tunnel release surgery.
* Steroid injection in carpal tunnel in the past 6 months.
* Cases of thoracic outlet syndrome and cervical radiculopathy.
* Pregnant females.
* Systemic rheumatic diseases such as rheumatoid arthritis.
* Hypothyroidism.
* Patients with bleeding tendency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-19 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 3 months post-procedure
  A visual analogue scale (VAS) via 11-point numerical pain rating scale (0=no pain to 10=maximum pain) was used to assess the current level of pain and hand discomfort

SECONDARY OUTCOMES:
Boston Questionnaire | 3 months post-procedure
  The Boston Questionnaire is a standardized, patient-based outcome measure of symptom severity and functional status in patients with carpal tunnel syndrome. The questionnaire including two parts, namely the symptom severity scales (SSS) and the functional status scales (FSS), is considered a standard tool to evaluate the patients with carpal tunnel syndrome (CTS). The SSS contains 11 questions on different symptoms of hand and FSS comprises of 5 questions assessing the difficulty in performing selected activities. The response to each question was scored from one (mildest) to five (most severe) points. The overall scores for SSS and FSS were calculated as the score sum of all questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.